CLINICAL TRIAL: NCT04708223
Title: A 24-Month Clinical Evaluation of an Ultra-rapid Polymerizing Resin Composite
Brief Title: Prospective, Split-mouth, Comparative Study to Compare Clinical Outcomes of Two Different Posterior Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LL3274680
Record Dates: First submitted 2020-12-22; First posted 2021-01-13 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-05

CONDITIONS: Caries; Defective Tooth Restorations

STUDY DESIGN:
Intervention Model Description: Split-mouth Design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fast-curing composites (Experimental)
  Interventions: Device: Direct restorative treatment with fast-curing composites (Tetric PowerFill/ Tetric PowerFlow)
- Conventionally applied composites (Other)
  Interventions: Device: Direct restorative treatment with conventionally applied composites (Tetric EvoCeram Bulk Fill/ Tetric EvoFlow Bulk Fill)

INTERVENTIONS:
Device: Direct restorative treatment with fast-curing composites (Tetric PowerFill/ Tetric PowerFlow) — Tooth (teeth) affected by dental caries or with an existing defective filling will be restored. Adhese Universal in self-etch mode, was used to prepare the surfaces for the composite fillings. Tetric PowerFill/ Tetric PowerFlow (test group) was cured for 3 s.
  Arms: Fast-curing composites
Device: Direct restorative treatment with conventionally applied composites (Tetric EvoCeram Bulk Fill/ Tetric EvoFlow Bulk Fill) — Tooth (teeth) affected by dental caries or with an existing defective filling will be restored. Adhese Universal in self-etch mode, was used to prepare the surfaces for the composite fillings. Tetric EvoCeram Bulk Fill/ Tetric EvoFlow Bulk Fill (control group) were conventionally cured for 10 s per increment.
  Arms: Conventionally applied composites

SUMMARY:
The objective of this 2-year split mouth comparative study, a randomized controlled study, is to determine whether the simplified placement procedure of the ultra-rapid polymerizing Tetric PowerFlow/ Tetric PowerFill with a reduced light polymerization time (3 s), yields the same clin-ical results as widely used commercially available dental composites (Tetric EvoCeram Bulk Fill, Tetric EvoFlow Bulk Fill) requiring up to 40 seconds of light polymerization time.

DETAILED DESCRIPTION:
Patients, requiring posterior tooth restorations Class I and II or requesting amalgam restoration replacement, were treated in the clinical investigation. Each patient received two composite restorations in the posterior region.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must need at least 2 restorations in a vital posterior tooth (in different quadrants)
* Restorations may be indicated for caries removal and restoration, replacement of defec-tive restorations (i.e. fractured, stained, unaesthetic), or requested replacement of un-aesthetic restorations.
* Must have given written consent to participate in the trial
* Must be available for the required follow-up visits over 2 years
* Restored teeth must have occlusal contact with opposing teeth or restored teeth
* Restoration width should be equal to or greater than 1/3 the distance from buccal to lin-gual cusp tips
* 75% of the restorations Class II (minimum) and 25% Class I
* One, two or three surfaces per restoration
* Each Class II will have at least one proximal contact
* 75% in molars (minimum) and 25% in premolars
* All restored teeth must have at least one occlusal contact in habitual closure
* Must have 20 or more teeth with evidence of bilateral posterior tooth contacts
* Teeth that require one or no cuspal build-ups
* Vital tooth
* Preoperative sensibility on the teeth to be treated at maximum 3 on visual analog scale (10 = maximum)
* Patient wishes to be treated in this clinical trial after oral information by the operator and after signing the informed patient form

Exclusion Criteria:

* Allergies to ingredients of the materials under investigation (monomers)
* Do not meet all inclusion criteria above
* Have medical complications (organ transplants, long term antibiotic or steroid treatment, cancer or are immunocompromised) or disabilities rendering them unable to tolerate the time required to complete the restorations or to provide adequate oral hygiene
* Suffer from xerostomia either by taking medications known to produce xerostomia or those with radiation induced xerostomia or Sjogren's syndrome subjects
* Have teeth with advanced or severe periodontitis, rampant caries or poor oral hygiene which may require extraction of the teeth to be restored
* Present with any systemic or local disorders that contraindicate the dental procedures included in this study
* Patients reporting having severe grinding/bruxing or clenching or in need of TMJ-related therapy
* Have tooth with exposed pulp during preparation or caries removal or require indirect pulp capping
* Inclusion of teeth that are non-vital or that exhibit signs of pulpal pathology (pulpitis)
* If the working field cannot be maintained in a dry state for treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon F. Cooper, Dr., Principal Investigator — University of Illinois College of Dentistry
Locations (1):
- University of Illinois College of Dentistry, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Teeth
Period: Overall Study
Arm/Group | Fast-curing composites | Conventionally applied composites
Started | 51; 50 Teeth | 51; 50 Teeth
6 Month | 49; 48 Teeth | 49; 48 Teeth
12 Month | 40; 36 Teeth | 40; 39 Teeth
24 Month | 37; 36 Teeth | 37; 37 Teeth
Completed | 31; 30 Teeth | 31; 29 Teeth
Not Completed | 20; 20 Teeth | 20; 21 Teeth

BASELINE CHARACTERISTICS:
Units Other Than Participants: Teeth
Groups:
- Total: Total of all reporting groups
Arm/Group | Fast-curing composites | Conventionally applied composites | Total
Number analyzed (Participants) | 51 | 51 | 153
Number analyzed (Teeth) | 50 | 50 | 100
Age, Customized [Number; unit: participants]
  number analyzed (Participants) | 51 | 51 | 51
  <= 18 years | 0 | 0 | 0
  18 to 80 years | 51 | 51 | 51
Sex/Gender, Customized [Number; unit: participants]
  number analyzed (Participants) | 51 | 51 | 51
  Female | 34 | 34 | 34
  Male | 17 | 17 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Teeth Analyzed According to FDI 11 - Postoperative Hypersensitivity
Description: assessed by tests with thermal stimuli and occlusal forces (during biting) determined by VAS (Visual Analog Scale, 0 "No pain at all" - 10 "The worst pain imaginable") following the Fédération dentaire internationale (FDI) criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: Baseline
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Fast-curing composites | Conventionally applied composites
Number analyzed (Participants) | 51 | 51
Number analyzed (Teeth) | 50 | 50
Teeth
  FDI 11 - Postoperative Hypersensitivity: FDI Score 1 | 47 | 45
  FDI 11 - Postoperative Hypersensitivity: FDI Score 2 | 3 | 5
  FDI 11 - Postoperative Hypersensitivity: FDI Score 3-5 | 0 | 0

2. Secondary Outcome: Restoration Quality Evaluation
Description: assessed following the FDI criteria (patient view, tooth vitality, surface luster, surface staining, colour match, material fracture, marginal adaption, occlusal wear and tooth integrity) on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: Baseline
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Fast-curing composites | Conventionally applied composites
Number analyzed (Participants) | 51 | 51
Number analyzed (Teeth) | 50 | 50
Teeth
  FDI 1 - Surface luster: FDI Score 1 | 44 | 41
  FDI 1 - Surface luster: FDI Score 2 | 6 | 9
  FDI 1 - Surface luster: FDI Score 3-5 | 0 | 0
  FDI 2 - Surface staining: FDI Score 1 | 50 | 47
  FDI 2 - Surface staining: FDI Score 2 | 0 | 3
  FDI 2 - Surface staining: FDI Score 3-5 | 0 | 0
  FDI 3 - Color match: FDI Score 1 | 28 | 24
  FDI 3 - Color match: FDI Score 2 | 20 | 19
  FDI 3 - Color match: FDI Score 3 | 2 | 7
  FDI 3 - Color match: FDI Score 4-5 | 0 | 0
  FDI 5 - Material fracture: FDI Score 1 | 50 | 49
  FDI 5 - Material fracture: FDI Score 2 | 0 | 1
  FDI 5 - Material fracture: FDI Score 3-5 | 0 | 0
  FDI 6 - Marginal adaption: FDI Score 1 | 49 | 49
  FDI 6 - Marginal adaption: FDI Score 2 | 1 | 0
  FDI 6 - Marginal adaption: FDI Score 3 | 0 | 0
  FDI 6 - Marginal adaption: FDI Score 4 | 0 | 1
  FDI 6 - Marginal adaption: FDI Score 5 | 0 | 0
  FDI 7 - Occlusal wear: FDI Score 1 | 50 | 50
  FDI 7 - Occlusal wear: FDI Score 2-5 | 0 | 0
  FDI 10 - Patient's view: FDI Score 1 | 39 | 42
  FDI 10 - Patient's view: FDI Score 2 | 8 | 4
  FDI 10 - Patient's view: FDI Score 3 | 3 | 2
  FDI 10 - Patient's view: FDI Score 4 | 0 | 2
  FDI 10 - Patient's view: FDI Score 5 | 0 | 0
  FDI 11 - Tooth vitality: FDI Score 1 | 50 | 50
  FDI 11 - Tooth vitality: FDI Score 2-5 | 0 | 0
  FDI 13 - Tooth integrity: FDI Score 1 | 50 | 48
  FDI 13 - Tooth integrity: FDI Score 2 | 0 | 2
  FDI 13 - Tooth integrity: FDI Score 3-5 | 0 | 0

3. Primary Outcome: Number of Teeth Analyzed According to FDI 11 - Postoperative Hypersensitivity
Description: assessed by tests with thermal stimuli and occlusal forces (during biting) determined by VAS (Visual Analog Scale, 0 "No pain at all" - 10 "The worst pain imaginable") following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 6 Month
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Fast-curing composites | Conventionally applied composites
Number analyzed (Participants) | 49 | 49
Number analyzed (Teeth) | 48 | 48
Teeth
  FDI 11 - Postoperative Hypersensitivity: FDI Score 1 | 46 | 47
  FDI 11 - Postoperative Hypersensitivity: FDI Score 2 | 1 | 1
  FDI 11 - Postoperative Hypersensitivity: FDI Score 3 | 1 | 0
  FDI 11 - Postoperative Hypersensitivity: FDI Score 4-5 | 0 | 0

4. Primary Outcome: Number of Teeth Analyzed According to FDI 11 - Postoperative Hypersensitivity
Description: as for outcome 3
Time Frame: 12 Month
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Fast-curing composites | Conventionally applied composites
Number analyzed (Participants) | 40 | 40
Number analyzed (Teeth) | 39 | 36
Teeth
  FDI 11 - Postoperative Hypersensitivity: FDI Score 1 | 38 | 36
  FDI 11 - Postoperative Hypersensitivity: FDI Score 2 | 1 | 0
  FDI 11 - Postoperative Hypersensitivity: FDI Score 3-5 | 0 | 0

5. Primary Outcome: Number of Teeth Analyzed According to FDI 11 - Postoperative Hypersensitivity
Description: as for outcome 3
Time Frame: 24 Month
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Fast-curing composites | Conventionally applied composites
Number analyzed (Participants) | 37 | 37
Number analyzed (Teeth) | 37 | 36
Teeth
  FDI 11 - Postoperative Hypersensitivity: FDI Score 1 | 36 | 36
  FDI 11 - Postoperative Hypersensitivity: FDI Score 2 | 1 | 0
  FDI 11 - Postoperative Hypersensitivity: FDI Score 3-5 | 0 | 0

6. Primary Outcome: Number of Teeth Analyzed According to FDI 11 - Postoperative Hypersensitivity
Description: as for outcome 3
Time Frame: 36 Month
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Fast-curing composites | Conventionally applied composites
Number analyzed (Participants) | 31 | 31
Number analyzed (Teeth) | 30 | 29
Teeth
  FDI 11 - Postoperative Hypersensitivity: FDI Score 1 | 30 | 28
  FDI 11 - Postoperative Hypersensitivity: FDI Score 2 | 0 | 0
  FDI 11 - Postoperative Hypersensitivity: FDI Score 3 | 0 | 1
  FDI 11 - Postoperative Hypersensitivity: FDI Score 4-5 | 0 | 0

7. Secondary Outcome: Restoration Quality Evaluation
Description: as for outcome 2
Time Frame: 6 Month
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Fast-curing composites | Conventionally applied composites
Number analyzed (Participants) | 49 | 49
Number analyzed (Teeth) | 48 | 48
Teeth
  FDI 1 - Surface luster: FDI Score 1 | 41 | 42
  FDI 1 - Surface luster: FDI Score 2 | 7 | 6
  FDI 1 - Surface luster: FDI Score 3-5 | 0 | 0
  FDI 2 - Surface staining: FDI Score 1 | 48 | 46
  FDI 2 - Surface staining: FDI Score 2 | 0 | 2
  FDI 2 - Surface staining: FDI Score 3-5 | 0 | 0
  FDI 3 - Color match: FDI Score 1 | 29 | 26
  FDI 3 - Color match: FDI Score 2 | 16 | 14
  FDI 3 - Color match: FDI Score 3 | 3 | 8
  FDI 3 - Color match: FDI Score 4-5 | 0 | 0
  FDI 5 - Material fracture: FDI Score 1 | 48 | 47
  FDI 5 - Material fracture: FDI Score 2 | 0 | 1
  FDI 5 - Material fracture: FDI Score 3-5 | 0 | 0
  FDI 6 - Marginal adaption: FDI Score 1 | 47 | 46
  FDI 6 - Marginal adaption: FDI Score 2 | 1 | 2
  FDI 6 - Marginal adaption: FDI Score 3-5 | 0 | 0
  FDI 7 - Occlusal wear: FDI Score 1 | 48 | 48
  FDI 7 - Occlusal wear: FDI Score 2-5 | 0 | 0
  FDI 10 - Patient's view: FDI Score 1 | 37 | 39
  FDI 10 - Patient's view: FDI Score 2 | 8 | 9
  FDI 10 - Patient's view: FDI Score 3 | 3 | 0
  FDI 10 - Patient's view: FDI Score 4-5 | 0 | 0
  FDI 11 - Tooth vitality: FDI Score 1 | 48 | 48
  FDI 11 - Tooth vitality: FDI Score 2-5 | 0 | 0
  FDI 13 - Tooth integrity: FDI Score 1 | 48 | 47
  FDI 13 - Tooth integrity: FDI Score 2 | 0 | 1
  FDI 13 - Tooth integrity: FDI Score 3-5 | 0 | 0

8. Secondary Outcome: Restoration Quality Evaluation
Description: as for outcome 2
Time Frame: 12 Month
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Fast-curing composites | Conventionally applied composites
Number analyzed (Participants) | 40 | 40
Number analyzed (Teeth) | 39 | 36
Teeth
  FDI 1 - Surface luster: FDI Score 1 | 35 | 32
  FDI 1 - Surface luster: FDI Score 2 | 4 | 4
  FDI 1 - Surface luster: FDI Score 3-5 | 0 | 0
  FDI 2 - Surface staining: FDI Score 1 | 36 | 29
  FDI 2 - Surface staining: FDI Score 2 | 2 | 5
  FDI 2 - Surface staining: FDI Score 3 | 1 | 2
  FDI 2 - Surface staining: FDI Score 4-5 | 0 | 0
  FDI 3 - Color match: FDI Score 1 | 17 | 17
  FDI 3 - Color match: FDI Score 2 | 18 | 18
  FDI 3 - Color match: FDI Score 3 | 4 | 1
  FDI 3 - Color match: FDI Score 4-5 | 0 | 0
  FDI 5 - Material fracture: FDI Score 1 | 38 | 36
  FDI 5 - Material fracture: FDI Score 2 | 1 | 0
  FDI 5 - Material fracture: FDI Score 3-5 | 0 | 0
  FDI 6 - Marginal adaption: FDI Score 1 | 36 | 33
  FDI 6 - Marginal adaption: FDI Score 2 | 3 | 2
  FDI 6 - Marginal adaption: FDI Score 3 | 0 | 0
  FDI 6 - Marginal adaption: FDI Score 4 | 0 | 1
  FDI 6 - Marginal adaption: FDI Score 5 | 0 | 0
  FDI 7 - Occlusal wear: FDI Score 1 | 39 | 36
  FDI 7 - Occlusal wear: FDI Score 2-5 | 0 | 0
  FDI 10 - Patient's view: FDI Score 1 | 33 | 30
  FDI 10 - Patient's view: FDI Score 2 | 4 | 5
  FDI 10 - Patient's view: FDI Score 3 | 2 | 1
  FDI 10 - Patient's view: FDI Score 4-5 | 0 | 0
  FDI 11 - Tooth vitality: FDI Score 1 | 39 | 36
  FDI 11 - Tooth vitality: FDI Score 2-5 | 0 | 0
  FDI 13 - Tooth integrity: FDI Score 1 | 36 | 34
  FDI 13 - Tooth integrity: FDI Score 2 | 2 | 2
  FDI 13 - Tooth integrity: FDI Score 3 | 1 | 0
  FDI 13 - Tooth integrity: FDI Score 4-5 | 0 | 0

9. Secondary Outcome: Restoration Quality Evaluation
Description: as for outcome 2
Time Frame: 24 Month
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Fast-curing composites | Conventionally applied composites
Number analyzed (Participants) | 37 | 37
Number analyzed (Teeth) | 37 | 36
Teeth
  FDI 1 - Surface luster: FDI Score 1 | 26 | 25
  FDI 1 - Surface luster: FDI Score 2 | 11 | 11
  FDI 1 - Surface luster: FDI Score 3-5 | 0 | 0
  FDI 2 - Surface staining: FDI Score 1 | 31 | 28
  FDI 2 - Surface staining: FDI Score 2 | 4 | 7
  FDI 2 - Surface staining: FDI Score 3 | 2 | 1
  FDI 2 - Surface staining: FDI Score 4-5 | 0 | 0
  FDI 3 - Color match: FDI Score 1 | 17 | 18
  FDI 3 - Color match: FDI Score 2 | 14 | 12
  FDI 3 - Color match: FDI Score 3 | 6 | 6
  FDI 3 - Color match: FDI Score 4-5 | 0 | 0
  FDI 5 - Material fracture: FDI Score 1 | 36 | 36
  FDI 5 - Material fracture: FDI Score 2 | 1 | 0
  FDI 5 - Material fracture: FDI Score 3-5 | 0 | 0
  FDI 6 - Marginal adaption: FDI Score 1 | 34 | 35
  FDI 6 - Marginal adaption: FDI Score 2 | 3 | 1
  FDI 6 - Marginal adaption: FDI Score 3-5 | 0 | 0
  FDI 7 - Occlusal wear: FDI Score 1 | 35 | 35
  FDI 7 - Occlusal wear: FDI Score 2 | 2 | 1
  FDI 7 - Occlusal wear: FDI Score 3-5 | 0 | 0
  FDI 10 - Patient's view: FDI Score 1 | 29 | 30
  FDI 10 - Patient's view: FDI Score 2 | 6 | 4
  FDI 10 - Patient's view: FDI Score 3 | 2 | 2
  FDI 10 - Patient's view: FDI Score 4-5 | 0 | 0
  FDI 11 - Tooth vitality: FDI Score 1 | 37 | 36
  FDI 11 - Tooth vitality: FDI Score 2-5 | 0 | 0
  FDI 13 - Tooth integrity: FDI Score 1 | 36 | 36
  FDI 13 - Tooth integrity: FDI Score 2 | 0 | 0
  FDI 13 - Tooth integrity: FDI Score 3 | 1 | 0
  FDI 13 - Tooth integrity: FDI Score 4-5 | 0 | 0

10. Secondary Outcome: Restoration Quality Evaluation
Description: as for outcome 2
Time Frame: 36 Month
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Fast-curing composites | Conventionally applied composites
Number analyzed (Participants) | 31 | 31
Number analyzed (Teeth) | 30 | 29
Teeth
  FDI 1 - Surface luster: FDI Score 1 | 20 | 20
  FDI 1 - Surface luster: FDI Score 2 | 10 | 9
  FDI 1 - Surface luster: FDI Score 3-5 | 0 | 0
  FDI 2 - Surface staining: FDI Score 1 | 26 | 20
  FDI 2 - Surface staining: FDI Score 2 | 4 | 9
  FDI 2 - Surface staining: FDI Score 3-5 | 0 | 0
  FDI 3 - Color match: FDI Score 1 | 15 | 13
  FDI 3 - Color match: FDI Score 2 | 8 | 10
  FDI 3 - Color match: FDI Score 3 | 7 | 6
  FDI 3 - Color match: FDI Score 4-5 | 0 | 0
  FDI 5 - Material fracture: FDI Score 1 | 30 | 29
  FDI 5 - Material fracture: FDI Score 2-5 | 0 | 0
  FDI 6 - Marginal adaption: FDI Score 1 | 28 | 25
  FDI 6 - Marginal adaption: FDI Score 2 | 2 | 4
  FDI 6 - Marginal adaption: FDI Score 3-5 | 0 | 0
  FDI 7 - Occlusal wear: FDI Score 1 | 30 | 29
  FDI 7 - Occlusal wear: FDI Score 2-5 | 0 | 0
  FDI 10 - Patient's view: FDI Score 1 | 26 | 25
  FDI 10 - Patient's view: FDI Score 2 | 3 | 3
  FDI 10 - Patient's view: FDI Score 3 | 1 | 1
  FDI 10 - Patient's view: FDI Score 4-5 | 0 | 0
  FDI 11 - Tooth vitality: FDI Score 1 | 30 | 29
  FDI 11 - Tooth vitality: FDI Score 2-5 | 0 | 0
  FDI 13 - Tooth integrity: FDI Score 1 | 27 | 24
  FDI 13 - Tooth integrity: FDI Score 2 | 0 | 2
  FDI 13 - Tooth integrity: FDI Score 3-5 | 0 | 0
  DI 13 - Tooth integrity: n/a | 3 | 3

ADVERSE EVENTS:
Time Frame: 36 Month
Arm/Group | Fast-curing composites | Conventionally applied composites
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 5/51 | 3/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fast-curing composites (N=51) | Conventionally applied composites (N=51)
Unrelated: Lesion next to study tooth (General disorders) | 1 | 0 — Patient showed sensitivity on study tooth due to a lesion on the tooth next to the study tooth
Buccal side repair (General disorders) | 0 | 1 — Buccal side repair due to material fracture
Unlikely related: Sensitivity near study tooth (General disorders) | 1 | 0
Sensitivity (General disorders) | 3 | 2 — It is generally related to this type of clinical procedure and might also be dependent on the applied light intensity, the used adhesive or the backstory of the tooth

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT04708223/Prot_SAP_001.pdf